CLINICAL TRIAL: NCT02132403
Title: PM-01: Phase 1b Study of PGG Beta Glucan (Imprime PGG®) in Combination With Anti-MUC1 Antibody (BTH1704) and Gemcitabine (Gemzar®) for the Treatment of Advanced Pancreatic Cancer
Brief Title: (PM-01) IMPRIME PGG® With BTH1704 and Gemcitabine for Advanced Pancreatic Cancer
Acronym: PM-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug Recall
Sponsor: University of Illinois at Chicago (Other)
Collaborators: HiberCell, Inc. (Industry)
Responsible Party: Principal Investigator, Howard Ozer, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1115
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; adenocarcinoma of the pancreas (PDAC); mixed adenocarcinoma of the pancreas; locally advanced; recurrent; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Anophthalmia with pulmonary hypoplasia; Recurrence; Neoplasm Metastasis | interventions — epitumomab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMPRIME PGG, BTH1704, & Gemcitabine (Experimental): Imprime PGG with BTH1704 at assigned doses administered on days 1, 8, 15, and 22 of a 28-day cycle with Gemcitabine on days 1, 8, and 15, at assigned doses, of a 28-day cycle.
  Interventions: Drug: BTH1704; Drug: IMPRIME PGG; Drug: Gemcitabine

INTERVENTIONS:
Drug: BTH1704 — BTH1704 at assigned doses administered on days 1, 8, 15, and 22 of a 28-day (4 week) cycle.
  Other Names: Humanized Human Milk Fat Globule 1 Antibody; huHMFG1; R1550; AS1402; Therex
Drug: IMPRIME PGG — Imprime PGG at assigned doses administered on days 1, 8, 15, and 22 of a 28-day (4 week) cycle.
  Other Names: Beta 1,3/1,6 glucan
Drug: Gemcitabine — Gemcitabine on days 1, 8, and 15, at assigned doses, of a 28-day (4 week) cycle.
  Other Names: Gemzar®

SUMMARY:
This Phase Ib dose escalation study will evaluate BTH1704, a monoclonal antibody that targets an aberrantly glycosylated antigen Mucin 1, and Imprime PGG, a glucan contained in yeast that is essential in triggering a leukocyte-mediated cytotoxic response towards tumor cells, in combination with gemcitabine in patients with advanced PDAC. The three intravenous drugs are taken in tandem 4 times in a 28-day cycle. The MAD of BTH1704 (BTH, 3 dose levels) in combination with gemcitabine (Gem) and Imprime PGG (I) will be determined using a standard "3+3" design. Treatment continues until disease progression, unacceptable toxicity, physician discretion, or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Histologically or cytologically confirmed adenocarcinoma of the pancreas, including pancreatic adenosquamous carcinoma, pancreatic anaplastic adenocarcinoma, pancreatic signet ring carcinoma, papillary mucinous carcinoma, acinar cell carcinoma, and ampulla of vater carcinoma,that is locally advanced (not able to proceed with surgery), recurrent, or metastatic (mixed adenocarcinoma of the pancreas is acceptable where the invasive component is predominantly adenocarcinoma)
3. Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1
4. Has an ECOG PS of 0, 1, or 2
5. Has been off chemotherapy for > or = 2 weeks
6. Has a patent biliary stent if required for biliary ductal obstruction, has adequate nutritional intake, and pain which is stable for a minimum of 24 hrs (pain score ≤ 3/10)
7. Has total bilirubin < 2 mg/dL, AST and ALT < 3.0 × ULN or < 5 x ULN for subjects with known hepatic metastases
8. Has serum creatinine < 2.5 × ULN
9. Has hemoglobin ≥ 9 g/dL, ANC ≥ 1.0 × 10^9/L, and platelet count ≥ 100 × 10^9/L
10. Must be willing and able to comply with study
11. Has read, understood and signed the ICF
12. Women of childbearing potential must not be pregnant or breast-feeding. In addition, a medically acceptable method of birth control must be used or total abstinence. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
13. Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male patients with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms at least 30 days after the last dose of study drug. Total abstinence is an acceptable alternative.
14. Prior systemic treatments for metastatic disease are permitted, including targeted therapies, biologic response modifiers, chemotherapy, hormonal therapy, or investigational therapy.
15. Availability of tissue if applicable (from the primary tumor or metastases)for banking
16. Willingness to donate blood for biomarker studies
17. Must have received at least one prior systemic chemotherapy on which disease progressed

Exclusion Criteria:

1. Has a diagnosis of resectable pancreatic adenocarcinoma
2. Had surgery within 4 weeks prior to study treatment
3. Has either untreated or symptomatic CNS mets
4. Has a known hypersensitivity to BTH1704, murine proteins, or any component of BTH1704
5. Has a known hypersensitivity to baker's yeast
6. Has had previous exposure to Imprime PGG
7. Has previously received an organ or progenitor/stem cell transplant
8. Has a history of blood clots, pulmonary embolism, or DVT unless controlled by anticoagulant treatment
9. Has a known history of HIV positivity or untreated & uncontrolled hepatitis B or C
10. Has any clinically significant infection
11. Has any other severe, uncontrolled medical condition, including uncontrolled DM or unstable CHF or has a known or suspected allergy to the study drug
12. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality that may increase the risk associated with study participation
13. Presence of any non-healing wound, fracture, or ulcer
14. Has any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance
15. Has any mental or medical condition that prevents the patient from giving informed consent
16. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to gemcitabine or drugs to formulate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 30 days post last dose
  The primary objective of this Phase 1b study is to determine the maximal administered dose (MAD) of BTH1704 (Mucin-1 targeted antibody) in combination with gemcitabine and Imprime PGG (beta 1,3/1,6 glucan) when given to patients with advanced and previously treated pancreatic ductal adenocarcinoma (PDAC).

SECONDARY OUTCOMES:
Adverse Effects | Up to 30 days post final dose
  Characterize adverse effects (AE) of I-BTH-Gem in patients with advanced PDAC in the second and third line setting.
Disease Response based on RECIST Criteria | Up to 8 weeks following final dose.
  Evaluate clinical response of I-BTH-Gem in patients with advanced PDAC in the second and third line setting (RECIST v 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Venepalli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UI Cancer Center, Chicago, Illinois, United States